CLINICAL TRIAL: NCT02318199
Title: Emergence Agitation During Recovery From Intracranial Surgery Under General Anesthesia: a Prospective Multicenter Cohort Study
Brief Title: Emergence Agitation in Adult Patients After Intracranial Surgery
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Municipal Administration of Hospital, China (Unknown)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY2014-034-01
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Intensive Care, Surgical; Postoperative Care; Neurosurgery
Keywords: emergence agitation; intracranial surgery; general anesthesia; incidence; risk factor
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Agitation group: Patient is evaluated by the sedation-agitation scale (SAS) during the anesthesia recovery after intracranial surgery under general anesthesia. SAS equals to 5-7 during the first 12 hours after surgery.
  Interventions: Procedure: Anesthesia recovery after intracranial surgery
- Non-agitation group: Patient is evaluated by the sedation-agitation scale (SAS) during the anesthesia recovery after intracranial surgery under general anesthesia. SAS equals to 1-4 during the first 12 hours after surgery.
  Interventions: Procedure: Anesthesia recovery after intracranial surgery

INTERVENTIONS:
Procedure: Anesthesia recovery after intracranial surgery — Intracranial surgery for brain tumor, traumatic brain injury, intracranial hemorrhage, subarachnoid hemorrhage and infection.

SUMMARY:
Emergence agitation is a frequent complication that can have serious consequences during recovery from general anesthesia. However, agitation has been poorly investigated in patients after craniotomy. In this prospective multicenter cohort study, adult patients will be enrolled after craniotomy and emergence agitation will be evaluated. The incidence, risk factors and outcome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Both supratentorial and infratentorial intradural cranial operations

Exclusion Criteria:

* Unarousable state (SAS=1) during the first 24 hours after the operation
* Interval longer than 24 hours between the end of the surgery and neurosurgical ICU admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients after craniotomy
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Emergence agitation | 12 hours after operation
  Emergence agitation is measured by sedation-agitation scale (SAS) and is defined as SAS=5-7.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (4):
- China (4):
  - Daxing Teaching Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Provincial Clinical College, Fujian Medical University, Fuzhou, Fujian
  - Bethune International Peace Hospital, Hebei Medical University, Shijiazhuang, Hebei
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia

REFERENCES:
- [Derived] Huang HW, Yan LM, Yang YL, He X, Sun XM, Wang YM, Zhang GB, Zhou JX. Bi-frontal pneumocephalus is an independent risk factor for early postoperative agitation in adult patients admitted to intensive care unit after elective craniotomy for brain tumor: A prospective cohort study. PLoS One. 2018 Jul 19;13(7):e0201064. doi: 10.1371/journal.pone.0201064. eCollection 2018. PMID 30024979
- [Derived] Yan LM, Chen H, Yu RG, Wang ZH, Zhou GH, Wang YJ, Zhang X, Xu M, Chen L, Zhou JX; Acute Brain Injury and Critical Care Research Collaboration (ABC Research Collaboration). Emergence agitation during recovery from intracranial surgery under general anaesthesia: a protocol and statistical analysis plan for a prospective multicentre cohort study. BMJ Open. 2015 Apr 21;5(4):e007542. doi: 10.1136/bmjopen-2014-007542. PMID 25900467